CLINICAL TRIAL: NCT04908631
Title: Safety and Feasibility of Transcranial Direct Current Stimulation to Enhance Auditory Rehabilitation in Cochlear Implant Recipients
Brief Title: Safety and Feasibility of tDCS to Enhance Auditory Rehabilitation in Cochlear Implant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00107525
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss
Keywords: Cochlear Implant
MeSH Terms: conditions — Hearing Loss | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- tDCS during auditory training (Other): Use of tDCS during completion of the auditory training program
  Interventions: Device: Transcranial Direct Stimulation; Other: Auditory Training Program

INTERVENTIONS:
Device: Transcranial Direct Stimulation — Brain stimulation using low-intensity current via electrodes on scalp to modify neuronal excitability in the underlying cortex. The tDCS system has customizable head gear with disposable, snap-in electrodes wihich can be applied at home without assistance.
  Other Names: tDCS 1x1 tES mini-CT, developed by Soterix Medical, USA
Other: Auditory Training Program — Web-based program uses consonant and vowel recognition and understanding sentences/conversations in quiet and in noise using different talkers, and other types of listening exercises.

SUMMARY:
This study aims to evaluate the safety and feasibility of transcranial direct current stimulation (tDCS) in combination with home-based auditory training therapy in cochlear implant (CI) patients. Changes in speech perception performance will also be evaluated.

DETAILED DESCRIPTION:
Participants will complete a 4 week web-based auditory training program while wearing a transcranial direct current stimulation device (tDCS). The customized auditory training program will be completed at home, in 20 - 30 minute sessions at least five times a week for four weeks. A customized learning and practice plan will be provided along with instructions on use of the tDCS device.

tDCS is a non-invasive brain stimulation technique that delivers low-intensity current via electrodes on the scalp to modify neuronal excitability in the underlying cortex. The tDCS system has customizable headgear with disposable, snap-in electrodes that are easy to apply at home without assistance.

Speech and hearing assessments will be completed prior to the start of auditory training, at the end of the 4 week training session, and again 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years of age
* Patients with a Unilateral Cochlear Implant device in use for a minimum of 1 year
* Sentence recognition scores (AzBio) below 65% and/or word recognition scores (CNC) are below 75% in the implanted ear for > one year following cochlear implantation.
* Ability to access internet to conduct computer-based auditory trainings and weekly video visits with study team weeks 2-5

Exclusion Criteria:

* Non-English speaking
* Diagnosis (documented or self-reported) of a psychiatric or neurologic condition, or any other comorbidities that may interfere with the study or increase the level of risk (such as dementia, seizures, legal blindness, brain tumor)
* Implants, other than CI, above collar bone level that may interact with delivery of tDCS
* Inability to or unwillingness to use electronic devices/computers, participate in video visits, or make required visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Francis, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | tDCS During Auditory Training
Started | 8
Completed | 5
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Received a second implant after the 1 month visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number Eligible Patients Who Expressed Interest in the Study
Time Frame: During the screening period of approximately 6 months
Population: Eligible patients who expressed interest in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 61
Participants | 61

2. Primary Outcome: Number of Subjects Who Completed tDCS Training
Description: Measured by total number of subjects enrolled who completed tDCS during auditory training
Time Frame: up to 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 8
Participants | 6

3. Primary Outcome: Number of Participants Who Demonstrated Competence of tDCS Training
Description: Measured by provider observation during in-office and tele-visits
Time Frame: 1 month
Population: One participant withdrew before the baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 7
Participants | 7

4. Primary Outcome: Number of Participants Who Reported Ease of Completing the Training Program
Description: Number of participants who reported agree or strongly agree as measured by questionnaire, where 1 equals strongly disagree and 5 equals strongly agree.
Time Frame: 1 month
Population: One participant withdrew before the baseline visit. One participant did not complete the training.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 6
Participants | 6

5. Primary Outcome: Number of Participants Who Reported an Adverse Event
Description: Measured by daily diary survey completion.
Time Frame: 30 days
Population: One participant withdrew before the baseline visit. One participant did not complete the daily diary.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 6
Participants | 0

6. Primary Outcome: Number of Participants Who Experienced Skin Irritation From Use of tDCS
Description: Measured by provider visual exam of scalp. Skin tingling/warmth is a known side effect of stimulation.
Time Frame: 6 months
Population: One participant withdrew before the baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 7
Participants | 6

7. Primary Outcome: Number of Subjects Who Experienced Abnormal Function of Cochlear Implant Device
Description: Measured by telemetry assessment.
Time Frame: 6 months
Population: One participant withdrew prior to the baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 7
Participants | 0

8. Primary Outcome: Speech Perception Performance - Sentence Recognition in Quiet
Description: Measured by word and sentence lists presented in quiet (AzBio Quiet). Average of two AzBio lists presented in quiet. Range of scores is from 0-100, with higher scores indicating higher speech perception performance.
Time Frame: Baseline, 1 month, 6 month
Population: Seven participants had a baseline assessment. One withdrew prior to 1 month; one additional participant withdrew prior to 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 7
score on a scale
  Baseline | 59.6 (33.1)
  1 Month: number analyzed (Participants) | 6
  1 Month | 68.8 (23.1)
  6 Months: number analyzed (Participants) | 5
  6 Months | 67.4 (25.4)

9. Primary Outcome: Speech Perception Performance - Word Recognition Performance
Description: Measured by 50-item CNC word list. CNC word lists are standardized sets of monosyllabic words used in audiology to assess speech recognition ability, particularly in cochlear implant users. Reported as a percentage (0-100%), with higher values indicating better word recognition.
Time Frame: Baseline, 1 month, 6 month
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of words
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 7
percentage of words
  Baseline | 43.1 (22.1)
  1 Month | 55.3 (21.9)
  6 Months | 47.2 (10.3)

10. Primary Outcome: Communication Function as Measured by Speech, Spatial and Qualities of Hearing (SSQ12) Questionnaire
Description: The SSQ12 questionnaire is scored as a mean of the 12 items, with a range of 0 to 10. A higher score indicates greater communication function.
Time Frame: Baseline, 1 month, 6 months
Population: One participant withdrew prior to 1 month; one additional participant withdrew prior to 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 7
score on a scale
  Baseline | 3.6 (1.9)
  1 month: number analyzed (Participants) | 6
  1 month | 4.5 (1.6)
  6 months: number analyzed (Participants) | 5
  6 months | 4.5 (2.1)

11. Primary Outcome: Cochlear Implant Quality of Life-35 Profile (CIQOL35) Questionnaire
Description: The CIQOL35 raw score is calculated by summing the items for each domain. In this case, the raw score for the Global 10 domain is reported. The range in raw scores is 10-50, where a higher score indicates great quality of life.
Time Frame: Baseline, 1 month, 6 months
Population: One participant withdrew prior to 1 month; one additional participant withdrew prior to 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 7
score on a scale
  Baseline | 32.9 (4.7)
  1 month: number analyzed (Participants) | 6
  1 month | 36.0 (6.1)
  6 months: number analyzed (Participants) | 5
  6 months | 36.8 (5.4)

12. Secondary Outcome: Number of Participants Who Enjoyed Doing the Listening Exercises on the Computer
Description: as for outcome 4
Time Frame: 1 month
Population: One participant withdrew before the baseline visit. One participant did not complete the training.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 6
Participants | 6

13. Secondary Outcome: Number of Participants Who Reported Use of the Stimulation Device to be Acceptable
Description: as for outcome 4
Time Frame: 1 month
Population: One participant withdrew before the baseline visit. One participant did not complete the training.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 6
Participants | 4

14. Secondary Outcome: Number of Participants Who Reported Improvement in Hearing Performance
Description: as for outcome 4
Time Frame: 1 month
Population: One participant withdrew before the baseline visit. One participant did not complete the training.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 6
Participants | 5

15. Secondary Outcome: Number of Participants Who Would Recommend the Training Program
Description: as for outcome 4
Time Frame: 1 month
Population: One participant withdrew before the baseline visit. One participant did not complete the training.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 6
Participants | 4

16. Secondary Outcome: Number of Participants Who Reported Acceptable Compensation for Study Participation
Description: as for outcome 4
Time Frame: 1 month
Population: One participant withdrew before the baseline visit. One participant did not complete the training.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS During Auditory Training
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: From the start of auditory training with tDCS at week 2 until the six-month follow-up visit
Description: Daily survey of known symptoms/side effects was submitted by the participant during training. One participant withdrew before the baseline visit.
Arm/Group | tDCS During Auditory Training
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT04908631/Prot_SAP_000.pdf